CLINICAL TRIAL: NCT05493345
Title: Active Communities - Adherence to Physical Activity Among Persons With Type 2 Diabetes, Cardiovascular Disease and/or Obesity - With a Focus on IT as a Tool
Brief Title: Active Communities - Adherence to Physical Activity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Steno Diabetes Center Sjaelland (Other Government); Center for Clinical Research and Prevention (Network)
Responsible Party: Principal Investigator, Mathias Ried-Larsen, Associate professor and Senior researcher, Rigshospitalet, Denmark
Other Study IDs: 21076311
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases; Obese
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Bridge-building between municipality-based lifestyle programs and community-based physical activities — Four co-created bridge-building activities has been implemented in the municipality of Odsherred, including (1) A digital portal for information and sharing of knowledge, (2) Visits between municipal rehabilitation programs and community-based physical activities, (3) Co-created teams for the target group, and (4) a 'Bridge builder' coordinator.

SUMMARY:
The primary aim of this study is to investigate whether a number of co-created bridge-building activities between municipality-based lifestyle programs and community-based physical activities (e.g. local sports and exercise associations) can support persons with type 2 diabetes, cardiovascular disease and/or obesity in maintain physical activity levels.

DETAILED DESCRIPTION:
This study is an evaluation of a number of co-created bridge-building activities between municipality-based lifestyle programs and community-based physical activities. Persons with type 2 diabetes, cardiovascular disease and/or obesity initiating a lifestyle program (8-12 weeks duration) in the municipality of Odsherred, Denmark, will be included in the study. We will include sixty (n=60) persons or the number of persons recruited at the end of the recruitment period, December 1, 2022 - whichever is reached first. Participants will undergo objective measurement of physical activity level, test of standing balance, 6-minute walk test, measurement of body composition, and answer questionnaires related to their background (education, job situation, civil status), health, lifestyle and well-being. Measurements will be performed before and after participants undergo a lifestyle program, and 3 and 6 months after termination of the lifestyle program.

ELIGIBILITY:
Inclusion Criteria:

* Citizens in the municipality of Odsherred undergoing a municipality-based lifestyle program
* Obese, or diagnosed with type 2 diabetes or cardiovascular disease

Exclusion Criteria:

* reliant on a wheelchair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Citizens with type 2 diabetes, cardiovascular disease and/or obesity in the municipality of Odsherred undergoing a municipality-based lifestyle program
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility and fidelity | From baseline (0 months) to follow-up (9 months)
  Feasibility and fidelity are evaluated using research progression criteria. Every domain is scored as either 1) Progress to RCT (randomized controlled trial) (green), 2) Amend before progressing to RCT (amber) or 3 do not progress to RCT (red).
  Domains include:
  * Satisfaction with project activities
  * Recruitment rate
  * Test- and participation burden
  * Retainment
  * Referral rate
  * Adherence
  * Physical activity improvement

SECONDARY OUTCOMES:
Moderate and vigorous physical activity (MVPA) time | From baseline (0 months) to follow-up (9 months)
  Change in time spend in MVPA (Accelerometer AX3)
Sitting time | From baseline (0 months) to follow-up (9 months)
  Change in time spend sitting (Accelerometer AX3)
Low-intensity physical activity (LPA) time | From baseline (0 months) to follow-up (9 months)
  Change in time spend in LPA (Accelerometer AX3)
Total physical activity (TPA) level | From baseline (0 months) to follow-up (9 months)
  Change in TPA measured in counts per minute (CPM) (Accelerometer AX3)
Steps | From baseline (0 months) to follow-up (9 months)
  Change in number of steps (Acceleromter AX3)
Six-minute walk distance | From baseline (0 months) to follow-up (9 months)
  Change in distance walked in a period of 6 minutes (6-minute walk test)
Standing balance | From baseline (0 months) to follow-up (9 months)
  Change in time spend in three standing positions (0-30 sec)
Body weight | From baseline (0 months) to follow-up (9 months)
  Change in body weight (bioimpedance scale)
Fat mass | From baseline (0 months) to follow-up (9 months)
  Change in fat mass (bioimpedance scale)
Fat percentage | From baseline (0 months) to follow-up (9 months)
  Change in fat percentage (bioimpedance scale)
Fat free mass | From baseline (0 months) to follow-up (9 months)
  Change in fat free mass (bioimpedance scale)
Muscle mass | From baseline (0 months) to follow-up (9 months)
  Change in muscle mass (bioimpedance scale)
Body mass index | From baseline (0 months) to follow-up (9 months)
  Change in body mass index (BMI)
Mental well-being | From baseline (0 months) to follow-up (9 months)
  Change in 5-item World Health Organization well-being index (WHO-5)
Risk of depression | From baseline (0 months) to follow-up (9 months)
  Change in number of participants scoring <50 in the WHO-5
Physical health-related quality of life | From baseline (0 months) to follow-up (9 months)
  Change in the SF-12 physical component summary (PCS)
Mental health-related quality of life | From baseline (0 months) to follow-up (9 months)
  Change in the SF-12 mental component summary (MCS)
Perceived stress | From baseline (0 months) to follow-up (9 months)
  Change in perceived stress scale (PSS) score
Loneliness | From baseline (0 months) to follow-up (9 months)
  Change in Three-Item Loneliness Scale (T-ILS) score

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Ried-Larsen, PhD, Principal Investigator — Centre for Physical Activity Research, Rigshospitalet
Locations (1):
- Centre for Physical Activity Research, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided